CLINICAL TRIAL: NCT03504735
Title: Effect of Caduet and TLC Intervention on Metabolic Parameters
Brief Title: Caduet and TLC Intervention in Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Pfizer (Industry); University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 082005-005
Record Dates: First submitted 2018-03-15; First posted 2018-04-20 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-04

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — amlodipine, atorvastatin drug combination; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Therapeutic Lifestyle Change+Placebo (Placebo Comparator): Therapeutic Life-style change intervention with Placebo pills.
  Interventions: Behavioral: Therapeutic Lifestyle Change; Drug: Placebo
- Therapeutic Lifestyle Change+Caduet (Active Comparator): Therapeutic Lifestyle Change intervention with Caduet pills.
  Interventions: Behavioral: Therapeutic Lifestyle Change; Drug: Caduet Pill

INTERVENTIONS:
Behavioral: Therapeutic Lifestyle Change — Monthly consult with a dietitian and fitness instructor.
  Other Names: TLC
Drug: Caduet Pill — Take once daily.
  Other Names: 5Mg-10Mg Tablet
  Arms: Therapeutic Lifestyle Change+Caduet
Drug: Placebo — Take once daily.
  Other Names: Oral Tablet
  Arms: Therapeutic Lifestyle Change+Placebo

SUMMARY:
To evaluate the effectiveness of Caduet in addition to therapeutic life-style change (TLC) intervention in resolving metabolic syndrome fifty three individuals were randomized to TLC intervention study with or without Caduet therapy for 12 months. The participants underwent monthly visits with investigators to obtain vital signs, and to undergo TLC counseling. Metabolic parameters were measured before and after intervention.

DETAILED DESCRIPTION:
Single center, investigator driven, double blinded, randomized with Caduet 5/10mg vs placebo. The participants visited with investigators on a monthly bases to evaluate the BP, weight, and obtain the waist measurements, and counseling. OGTT was performed at the beginning and the end of the study. Lipid and glucose parameters were measured 5 times in duration of the study period.

Exercise physiologists and dietitians completed the baseline evaluations and provided recommendations throughout the study period in person, via phone or e-mail: per subject preference. VO2 max was measured at the beginning and end of the study. Pedometers dispensed to encourage physical activity.

ELIGIBILITY:
Inclusion Criteria:

* BP ≥130/85
* Metabolic syndrome per NCEP-ATP III revised (3/5 criteria)
* Men and women age 40-65

Exclusion Criteria:

* Inability to sign a consent form.
* Unwillingness to complete the protocol for the duration of 15 months
* Unwillingness of primary care physician to participate in the program
* Patients already on hypercholesterolemia agent
* Fasting plasma glucose above 126 mg/dL or current treatment for diabetes.
* If the physician believes the patient should be started on antihypertensive regimen.
* Creatinine clearance <50ml/min.
* Therapy with anticoagulants
* Pregnant/lactating women (pre-menopausal women should be on birth control pill)
* AST/ALT > x3 upper limit of normal
* Evidence of cholelithiasis
* Use of oral anticoagulants
* Cancer
* Recent cardiovascular event (<6months)
* Substance abuse
* Since there is no translator, non-English speaking subjects will not be enrolled in the study.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2005-05-01 (Actual); Primary Completion 2009-01-01 (Actual); Study Completion 2016-02-28 (Actual)

PRIMARY OUTCOMES:
Resolution or improvement of metabolic syndrome. | 12 months
  HDL >40mg/dl for men, >50 mg/dl for women. Glucose <100mg/dl Waist circumference <40 in in men, <35 in in women Triglycerides <150mg/dl BP <130/80 Attainment of 1 or more of these goals will result in resolution or improvement of metabolic syndrome

SECONDARY OUTCOMES:
Weight loss | 12 months
  5% decrease compared to that at the start of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Abate, MD, Principal Investigator — University of Texas

IPD SHARING:
Plan to Share IPD: No